CLINICAL TRIAL: NCT00220077
Title: Determination of the Role of Microarray for Prognosis and Prediction to Chemotherapy Sensitivity in Patients With Operable, Locally Advanced and Metastatic Oesophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2110
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Oesophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Endoscopy

INTERVENTIONS:
Procedure: Endoscopy

SUMMARY:
Knowledge of the impact of gene expression profiling could allow optimisation of chemotherapy regimens for individual patients. It could ensure that patients do not receive a particular form of chemotherapy if it is unlikely to benefit them, and in these circumstances an alternative form of chemotherapy that may prove beneficial could be selected. This information will therefore allow chemotherapy to be tailored to the individual tumour. It may help identify those patients with a poorer prognosis who could be selected for further therapy post surgery or a different treatment strategy at the outset.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with histologically proven operable ,locally advanced and metastatic oesophageal or gastric carcinoma.

Exclusion Criteria:

* Second malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2002-06

PRIMARY OUTCOMES:
To determine whether specific gene expression profiles are associated with response in oesophago-gastric cancer.

SECONDARY OUTCOMES:
Evaluation of the association of gene expression profiling and progression free survival and overall survival in patients with oesophago-gastric cancer.

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom